CLINICAL TRIAL: NCT00270569
Title: A Phase II Study of Weekly Low-Dose Paclitaxel Plus 24-Hour Infusion of Cisplatin as First-Line Chemotherapy for Metastatic Breast Cancer
Brief Title: An Effective and Compliance Regimen of Paclitaxel Plus Cisplatin to Treat Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Far Eastern Memorial Hospital, Far Eastern Memorial Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FEMH-94012
Record Dates: First submitted 2005-12-26; First posted 2005-12-28 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2005-08

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Cisplatin

INTERVENTIONS:
Drug: PhyxolTM, Cisplatin

SUMMARY:
The primary endpoint of this phase II trial is the objective response rate of the stage I (low-dose) regimen. The secondary endpoints include treatment-related toxicity, the change in quality of life, progression free survival and overall survival. Simon's optimal two-stage design will be used to determine the patient number.

DETAILED DESCRIPTION:
Breast cancer is one of the leading causes of cancer death for women in Taiwan. We have recently demonstrated that combination of paclitaxel and cisplatin, at conventional doses, is highly effective in the treatment of breast cancer. However, the acute and cumulative toxicities of paclitaxel have been troublesome to a significant portion of the patients. Several lines of evidence suggested that weekly paclitaxel, at a much lower dose range of 40 to 50 mg/m2 per week, may be as effective as that of the conventional doses of paclitaxel (80 to 90 mg/m2 per week) for patients with metastatic ovarian and lung cancers. The low-dose regimen of paclitaxel may significantly improve the compliance of the patients. This open-label phase II trial is designed to test this hypothesis.

The eligibility criteria include (1) women with metastatic breast cancer; (2) measurable disease; (3) acceptable organ function reserves. The ineligibility criteria include (1) brain or leptomeningeal metastases; (2) previous chemotherapy for metastatic breast cancer. The study consists of two stages. All eligible patients will receive stage I (low-dose) regimen: paclitaxel, 50 mg/m2 1-hour iv infusion on days 1, 8 and 15, and cisplatin, 40 mg/m2 24-hour iv infusion on days 1 and 8. The treatment cycle will be repeated every 4 weeks. The first tumor response assessment will be done after 2 cycles of protocol treatment. Patients with complete response (CR) will receive at least 2 more cycles of low-dose regimen after documentation of CR. Patients with partial response (PR) and patients with stable disease (SD) who have minor tumor response or improvement of general condition will continue to receive the low-dose regimen. Patients with SD but no evident clinical benefit and patients with progressive disease (PD) will be shifted to stage II (conventional-dose) regimen: paclitaxel, 80 mg/m2 1-hour intravenous infusion on days 1, 8 and 15, and cisplatin, 40 mg/m2 24-hour intravenous infusion on days 1 and 8, every 4 weeks. Tumor assessment will then be evaluated after every 2 cycles of protocol treatment. For patients who continue low-dose regimen, those with CR will receive at least 2 more cycles of protocol treatment. Patients with a maximal response of PR or SD may either continue the low-dose regimen until PD or prohibitive toxicity develops or change to the conventional-dose regimen, at the discretion of the attending physicians. Patients with PD should change to the conventional-dose regimen. For patients who have shifted to conventional-dose regimen, those with CR will receive at least 2 more cycles of protocol treatment. Patients with PR will continue protocol treatment until disease progresses or prohibitive toxicity develops. Patients with SD may continue protocol treatment or change to salvage therapy. Patients with PD should stop protocol treatment and change to salvage therapy.

The primary endpoint of this phase II trial is the objective response rate of the stage I (low-dose) regimen. The secondary endpoints include treatment-related toxicity, the change in quality of life, progression free survival and overall survival. Simon's optimal two-stage design will be used to determine the patient number. If 4 or more objective responses (CR+PR) are documented in the first 13 patients, the study will go on to the second stage to enroll a total of 43 patients. The P0, P1,are 20%, 40%, 0.05, and 0.2, respectively. Assuming a dropout rate of 10%, 15 patients will be accrued in the first stage and 33 in the second stage. Estimated time for patient accrual is 3 years.

ELIGIBILITY:
Inclusion Criteria:

* 1.Women with histologically proven breast cancer and clinical evidence of distant metastasis. (AJCC staging, 2002; see Appendix I)
* 2.Bi-dimensionally measurable disease by physical examination or image study (roentgenogram or computed tomography (CT) scan). The index lesions should be at least 20 mm × 20 mm in size.
* 3.Age must be older than 18 and younger than 75 year-old.
* 4.Karnofsky performance status 70%. (see Appendix)
* 5.Adequate bone marrow reserves, defined as white blood cell(WBC)4,000/l, absolute neutrophil count (ANC) 1,500/l, platelet 100,000/l.
* 6.Liver transaminases 3 times upper normal limit if no liver metastasis and 5 times upper normal limit if liver metastasis is present; total bilirubin 2 mg/dl;serum creatinine 1.5 mg/dl.
* 7.No prior chemotherapy for metastatic disease. Previous chemotherapy as adjuvant treatment is acceptable, if the adjuvant chemotherapy has been completed at least 6 months before entry into in this study.
* 8.If the patients have received hormonal therapy for metastatic disease, there must be definite evidence of disease progression under the hormonal therapy,and hormonal therapy should be discontinued before entry into this study.
* 9.Previous or concurrent radiotherapy is acceptable if the area of radiation does not involve the site of the index tumor lesions.
* 10.Patients of childbearing age should have effective contraception during the study period.
* 11.All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional guidelines.

Exclusion Criteria:

* 1.Patients who are receiving concurrent hormonal or cytotoxic therapy or other experimental therapy.Concurrent therapy with other biological agents, such as Trastuzumab (Herceptin), is not allowed.
* 2.Patients who refuse port-A catheter implantation.
* 3.Patients who have received taxane (paclitaxel or docetaxel) or cisplatin as adjuvant chemotherapy.
* 4.Patients with brain or leptomeningeal metastases.
* 5.Patients who have significant cardiac arrhythmia or acute myocardial infarction within 6 months before entry.
* 6.Patients who have major systemic diseases that the attending physicians considered inappropriate for systemic chemotherapy.
* 7.Life expectancy less than 2 months.
* 8.Pregnant or nursing patients may not participate. Patients with reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
* 9.No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancers, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any cancer from which the patient has been disease-free for 5 years.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2005-10; Primary Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
The primary objective is to determine the tumor response of weekly low-dose paclitaxel plus 24-hour infusion of cisplatin chemotherapy for patients with metastatic breast cancer.

SECONDARY OUTCOMES:
Toxicities of weekly low- or conventional-dose paclitaxel plus 24-hour infusion of cisplatin.
The patients'quality of life as evaluated by questionnaire interview.
Progression-free survival.
Overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Kun Huei Yeh, Ph.D., Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, Taipei, Ban-Ciao, Taiwan